CLINICAL TRIAL: NCT01129570
Title: Phase I Trial of Siliphos in Patients With Advanced Hepatocellular Carcinoma
Brief Title: Siliphos in Advanced Hepatocellular Carcinoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Abby Siegel (Other)
Collaborators: Lotte & John Hecht Memorial Foundation (Other)
Responsible Party: Sponsor-Investigator, Abby Siegel, Assistant Professor of Clinical Medicine, Oncology, Columbia University
Organization: Columbia University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAE7604
Record Dates: First submitted 2010-04-12; First posted 2010-05-24 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-11

CONDITIONS: Advanced Hepatocellular Carcinoma
MeSH Terms: interventions — Silybin; milk-thistle extract; TXNIP protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Siliphos - dose escalation (Experimental)
  Interventions: Drug: Silybin

INTERVENTIONS:
Drug: Silybin — 4 dose levels of siliphos: 2, 4, 8, and 12 grams daily in three divided doses. This study will follow a standard sequential Phase I dose escalation design.
  Other Names: Siliphos; Milk thistle; Advanced hepatocellular carcinoma

SUMMARY:
Milk thistle is an herbal drug that may have some liver protection properties and may reduce inflammation in the liver. It may also have anticancer effects. However milk thistle is not approved by the Food and Drug Administration for any medical purpose in the United States.

It has not been used in patients with liver cancer previously, to our knowledge, but there have been many studies of its use in patients with hepatitis and cirrhosis. Some of these studies have shown that milk thistle may help reduce elevated liver function tests.

Siliphos is a derivative of milk thistle that can be absorbed better than some other types of milk thistle. The investigators would like to perform a study to identify doses of siliphos that are safe to take in advanced liver cancer and to identify positive or negative side effects this compound may have. The investigators will be using this information in future studies to see if siliphos can be used as a therapy in patients with advanced liver cancer to reduce elevated liver function tests.

DETAILED DESCRIPTION:
Milk thistle (MT) has been historically used to treat patients with liver diseases, and has been shown to have antioxidant, anti inflammatory, and hepatoprotective properties. It may also have direct anticancer effects through inhibition of growth factors and promotion of cell cycle arrest. MT has been shown to improve LFTs in several studies of patients with cirrhosis. To our knowledge, there have been no published trials evaluating the clinical efficacy of MT in advanced HCC. We therefore propose a phase I study to identify the maximum tolerated dose (MTD) of silybinphosphatidylcholine (a commercially available preparation with increased bioavailability), in patients with advanced HCC. We will use a traditional dose escalation, open label design with a study intervention period of 3 months, followed by one year of observation, with a maximum total of 30 subjects, evaluating a dose range between 1 to 12 gm Siliphos. The data obtained from this study will be utilized in the future to evaluate MT efficacy in reducing liver function tests in advanced HCC, which will have significant implications in its use as a potential adjunctive agent in patients with currently limited treatment options.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* ECOG performance score of 0-3
* Expected survival of >12 weeks
* Subjects with advanced HCC or locally advanced, unresectable HCC
* Elevated LFTs (including at least one of the following: TBili >1.5 times the upper limit of normal; serum AST >2.5 times the upper limit of normal
* HCC diagnosed/defined based on either biopsy, or by suggestive radiologic imaging according to the AASLD guidelines (arterial enhancement with venous washout) or an AFP >200 ng/ml
* Subjects must have measurable disease that can be accurately measured in at least one dimension (with at least >20mm diameter in the longest dimension by conventional imaging or >10 mm by helical CT)
* Elevated liver enzymes that are either due to underlying liver disease and/or tumor which is not amenable to stenting after discussion with interventional GI and/or IR
* Subjects must demonstrate an ability to understand the consent process and willingness to sign a written informed consent form
* Subjects must agree to use birth control pills or other active contraception during active study treatment

Exclusion Criteria:

* Pregnant women or women currently breastfeeding will be excluded from this study because the effects of silybin on pregnant women and/or nursing infants are not known
* Subjects must have < grade 4 hepatic toxicity
* Known brain metastases because of poor prognosis and as patients with brain metastases often develop neurological dysfunction that may confound evaluation of neurologic and other adverse side effects
* History of allergic reactions to the study medication
* Uncontrolled concurrent illness including, but not limited to: ongoing active infection (including SBP), symptomatic congestive heart failure, unstable angina, active cardiac arrhythmia, or psychiatric illness that would limit compliance with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2010-02; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
The maximum tolerated dose of siliphos in patients with advanced hepatocellular carcinoma | Weeks 1, 3, 6, 9, and 12

SECONDARY OUTCOMES:
Mean intra-patient percent change in AST, ALT and total serum bilirubin levels | From baseline to 3 months
  Fasting morning blood samples collected at baseline, weeks 1, 3, 6, 9, and 12
Quality of life as measured by the FACT-hepatobiliary questionnaire | From baseline to 3 months
  Questionnaire administered at baseline, weeks 1, 6, and 12
Plasma concentrations of silybinin, silybinin B, silibinin glucoronide, and silibinin sulfate | From baseline to 3 months
  Fasting morning blood samples collected at baseline, weeks 1, 3, 6, 9, and 12
Mean intra-patient percent change in serum concentrations of CRP, IGF-1, and IGFBP-3 | From baseline to 3 months
  Fasting morning blood samples collected at baseline, weeks 1, 3, 6, and 12
Tumor response as measured by RECIST criteria and AFP concentrations | From baseline to 3 months
  Fasting blood samples collected at baseline, weeks 1, 3, 6, 9, and 12 for AFP concentrations.
  MRI of abdomen/pelvis & CT of chest at baseline and week 12

CONTACTS AND LOCATIONS:
Overall Officials: Abby Siegel, MD, MS, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States